CLINICAL TRIAL: NCT00198406
Title: A FRENCH SURVEY OF THE DIAGNOSTIC AND THERAPEUTIC MANAGEMENT OF ELDERLY PEOPLE WITH HISTOLOGICALLY/CYTOLOGICALLY CONFIRMED LUNG CANCER.
Status: Completed | Type: Observational
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Other Study IDs: IFCT-0202
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: ELDERLY PEOPLE; Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: diagnostic and therapeutic management

SUMMARY:
Management of lung cancer remains very controversial for elderly patients (pts) and they are often excluded from clinical trials. We present here a survey performed about the management of lung cancer pts aged 70 or more in France. All pts aged 70 or more with histo/cytologically proved lung cancer diagnosed between sept 02 and oct 03 in participating centers were recorded and their characteristics, the diagnostic procedures, therapeutic management and survival were analysed.

ELIGIBILITY:
Inclusion Criteria:

* histo/cytologically proved lung cancer

Exclusion Criteria:

-

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1653
Dates: Start 2002-09; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Quoix, Principal Investigator — Intergroupe Francophone de Cancerologie Thoracique
Locations (1):
- CHU Lyautey - Pneumologie, Strasbourg, France